CLINICAL TRIAL: NCT06200259
Title: Reduction of Gastrointestinal Toxicity in Prostate Cancer by Proton Spot Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Covenant Health Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-485 INV
Record Dates: First submitted 2023-12-13; First posted 2024-01-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- "Spot Delete" (Experimental): A unique technique called "Spot Delete" will be utilized to control the placement of spots during treatment planning, to prohibit proton spots from being placed in the rectum, sigmoid, and small bowel. A specialized computer model will be used to study how the energy of the proton beam (linear energy transfer) is related to rectal and bladder side effects.
  Interventions: Radiation: Spot Delete planning for proton therapy
- Control Arm (Active Comparator): The proton spots that are placed by the treatment planning system are not modified
  Interventions: Radiation: Traditional proton treatment planning system

INTERVENTIONS:
Radiation: Spot Delete planning for proton therapy — The method of adjusting the placement of proton spots or targets that are placed by the treatment planning system during pencil beam scanning for proton therapy
  Other Names: Pencil beam scanning proton therapy
  Arms: "Spot Delete"
Radiation: Traditional proton treatment planning system — In the control arm, the proton spots placed by the treatment planning system are not modified.
  Arms: Control Arm

SUMMARY:
This purpose of this study is to examine the placement of proton spots during pencil beam scanning proton therapy for low and intermediate risk prostate cancer. The researchers will test a unique technique called "Spot Delete" to control the placement of spots during treatment planning. They will also use a special computer model to study how the energy of the proton beam (linear energy transfer) is related to rectal and bladder side effects. The study involves creating a treatment plan based on a CT scan, which helps guide the proton beam in the body. The clinical team uses this CT scan to find the best placement for the protons. The "Spot Delete" method prevents protons from stopping in the rectum, sigmoid, and small bowel, which is thought to be related to acute or late toxicities, such as tenesmus, diarrhea, fecal incontinence, proctitis, and rectal hemorrhage.

DETAILED DESCRIPTION:
Patients will be randomized into two groups of spot placement. In the experimental arm, "Spot Delete" will be used to prohibit proton spots from being placed in the rectum, sigmoid, and small bowel. In the control arm, proton spots are placed by the treatment planning system are not modified. Medical staff will document gastrointestinal toxicities (diarrhea, fecal incontinence, proctitis, and rectal hemorrhage) and genitourinary toxicities (hematuria, urinary incontinence, urinary retention, urinary obstruction, urinary pain, urinary frequency, and urinary urgency) in the electronic medical record.

This study carries the same risks as regular proton therapy. Proton therapy, like other cancer treatments, may cause the aforementioned side effects. It is important to note that the "Spot Delete" technique aims to specifically address the bladder and bowel reactions, so there might be a potential reduction in this particular risk. Dose constraints will be the same for each treatment arm. Though not expected, it is theoretically possible that this method may counterintuitively increase side effects involving the bladder or bowel. Likewise, increased side effects in other organs are not expected, but are theoretically possible. For this reason we believe there is clinical equipoise between the two trial arms.

ELIGIBILITY:
Inclusion Criteria:

* Pathological proven diagnosis of prostatic adenocarcinoma
* History and physical exam to establish clinical staging
* Clinical stage T1-T2c (AJCC 7th edition)
* Prostate specific antigen (PSA) < 20 ng/mL
* Gleason Score ≤ 7
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-1
* Patients must be 18 years of age or older
* Willingness and ability to complete the International Prostate Symptom Score (IPSS) survey and Expanded Prostate Cancer Index Composite (EPIC) questionnaire

Exclusion Criteria:

* Prior radiotherapy to the pelvic area
* Prior prostate cancer therapy: cryotherapy or hyperthermia
* Prior systemic therapy (chemotherapy) for prostate cancer
* Regional lymph nodes (common iliac, external iliac, internal iliac, presacral) are a target of treatment
* Active diverticulitis, ulcerative colitis, or Crohn's disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pathological proven diagnosis of prostatic adenocarcinoma
Enrollment: 500 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2040-01-02 (Estimated)

PRIMARY OUTCOMES:
Test the hypothesis that "Spot Delete" technique in proton therapy reduces late toxicity in low- and intermediate-risk prostate cancer patients | assessed at baseline, during treatment, at the end of treatment, and annually up to 10 years
  The effectiveness of the technique will be evaluated by measuring and documenting the degree of GI and GU reactions in patients undergoing proton therapy with the "Spot Delete" technique. Diarrhea, Fecal Incontinence, Proctitis, Rectal Hemorrhage, Hematuria, Urinary Incontinence, Urinary Retention, Urinary Obstruction, Urinary Pain, Urinary Frequency, and Urinary Urgency will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) ver. 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Hedrick, PhD, DABR, Principal Investigator — Thompson Proton Center
Locations (1):
- Thompson Proton Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No